CLINICAL TRIAL: NCT05844163
Title: Treatment Strategies for Unruptured Intracranial Aneurysms in the Chinese Population China Treatment Trial for Unruptured Intracranial Aneurysm (ChTUIA)
Acronym: ChTUIA
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Huashan Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Fujian Medical University (Other); Shanxi Provincial People's Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Shuo, Director of Department of Cerebrovascular Neurosurgery, Beijing Tiantan Hospital
Other Study IDs: KY2022-226
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-11

CONDITIONS: Unruptured Intracranial Aneurysm
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Intracranial aneurysm clipping group: Patients in Intracranial aneurysm clipping group receive neurosurgical clipping.
  Interventions: Other: observation
- Coil embolization or stent-assisted coil embolization group: Patients in coil embolization or stent-assisted coil embolization group receive coil embolization or stent-assisted coil embolization according to individualized condition.
  Interventions: Other: observation
- Flow diversion group.: Patients in flow diversion group receive flow diverters.
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — observation

SUMMARY:
The goal of this prospective observational cohort study is to learn about treatment strategies for unruptured intracranial aneurysms in the Chinese population. The main questions it aims to answer are:

* To establish a cohort of patients with intracranial unruptured aneurysm and explore the optimal clinical treatment strategy.
* To establish clinical management path for patients with unruptured intracranial aneurysm.

According to the treatment of all patients with unruptured intracranial aneurysm, they were divided into the following groups: 1. Conservative treatment group; 2. Intracranial aneurysm clipping group; 3. Coil embolization or stent-assisted coil embolization group; 4. Flow diversion group.

ELIGIBILITY:
Inclusion Criteria:

A. age > 18 years. B. at least one intracranial aneurysm needs to be treated by craniotomy, endovascular treatment or combined surgery.

C. patients' consent were obtained.

Exclusion Criteria:

1. Ruptured intracranial aneurysms, accompanied by subarachnoid hemorrhage or cerebral hemorrhage ;
2. Traumatic, infectious and atrial myxoma-associated intracranial aneurysms ;
3. Combined with cerebrovascular malformations;
4. Combined with brain tumors or malignant tumors in other parts ;
5. Combined with systemic connective tissue disease and systemic rheumatic disease ;
6. Due to other diseases, or poor general condition, the expected survival time is not more than 12 months ;
7. During pregnancy and perinatal period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unruptured intracranial aneurysm
Sampling Method: Probability Sample
Enrollment: 31595 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | 2 years
  Functional outcomes(modified Rankin Scale,mRS) at 2 years after treatment decision

SECONDARY OUTCOMES:
MACCE events | 1 years
  Incidence of major adverse cardiovascular/cerebrovascular events (MACCE events) in patients with atherosclerotic heart disease within 1 year after treatment decision.
cardiovascular/cerebrovascular events | 2 years
  Incidence of cardiovascular/cerebrovascular events in 2 years after receiving different treatment strategies.
Cost | 2 years
  Costs associated with unruptured intracranial aneurysms within 2 years after treatment with different strategies.
Aneurysm-related bleeding events | 2 years
  Incidence of aneurysmal-related bleeding events within 2 years after receiving different treatment strategies.
Mortality associated with intracranial aneurysms | 2 years
  Mortality associated with intracranial aneurysms within 2 years after treatment with different strategies
All-cause mortality | 2 years
  All-cause mortality of patients within 2 years after different treatment strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Wang shuo, M.D., Study Chair — Beijing Tiantan Hospital
Locations (1):
- Capital Medical University Affiliated Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng K, Wen Z, Wang K, Mo S, Wu J, Chen X, Zhao B, Liu Q, Wang S. Treatment strategies for unruptured intracranial aneurysms in the Chinese population: China Treatment Trial for Unruptured Intracranial Aneurysm (ChTUIA). Chin Neurosurg J. 2025 Apr 3;11(1):8. doi: 10.1186/s41016-025-00394-7. PMID 40181400